CLINICAL TRIAL: NCT02871856
Title: International Lung Screen Trial
Brief Title: International Lung Screen Trial (ILST)
Acronym: ILST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, Kwun Fong, Professor, The University of Queensland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HREC/16/QPCH/181
Record Dates: First submitted 2016-08-08; First posted 2016-08-18 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Smokers at Risk of Lung Cancer
Keywords: Screening; Computed tomography; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Other): Single arm only, CT screening of lung
  Interventions: Diagnostic Test: Low dose CT

INTERVENTIONS:
Diagnostic Test: Low dose CT — low-dose screening CT of chest for lung cancer detection

SUMMARY:
People who may be at increased risk of lung cancer due to age and smoking history will be invited to participate in this international study to determine the best way of using computed tomography (CT) of the chest to screen for early lung cancer. Overseas data show that CT screening (screening tests can find diseases early, when they're easier to treat) can reduce deaths from lung cancer and this study will help determine who is most likely benefit from screening.

DETAILED DESCRIPTION:
[insert site name]

ELIGIBILITY:
* Inclusion Criteria:
* Women or men age from 55 to 80.
* Current or former smokers. A former smoker is defined as one who has stopped smoking for one or more years.
* An estimated 6-year lung cancer risk of ≥1.51% based on the PLCOm2012 risk prediction model or ≥ 30 pack-years smoking history (pack-year is defined as number of pack of cigarettes smoked per day multiply by the number of years smoked. If a participant stopped smoking for 6 months or more and then restarted smoking again, the time will be subtracted from the total duration of smoking in 0.5 year increments)
* ECOG performance status 0 or 1.
* Capable of providing, informed consent for screening procedures (low dose spiral CT)
* Exclusion Criteria
* Clinical symptoms suspicious for lung cancer e.g. hemoptysis, chest pain, weight loss
* Any medical condition, such as severe heart disease (e.g. unstable angina, chronic congestive heart failure), acute or chronic respiratory failure, home oxygen therapy, bleeding disorder, that in the opinion of the investigator could jeopardize the subject's safety during participation in the study or unlikely to benefit from screening due to shortened life-expectancy from the co-morbidities
* Have been previously diagnosed with lung cancer
* Have had other non-curatively treated cancer outside the lung.
* Pregnancy
* Pneumonia or bronchitis requiring antibiotic treatment within the last 12 weeks
* Unwilling to have a spiral chest CT
* Chest CT within 2 years
* Does not fit into CT scanner table due to gross obesity
* Cannot lie on CT scanning table on the back with arms over the head
* Received chemotherapy or cytotoxic drugs within the last 6 months
* Unwilling to sign a consent

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The number of Lung cancers | 5 years
Number of nodules | 5 years
Change in quality of life | 5 Years

SECONDARY OUTCOMES:
Cancer detection rate | 5 years
Types and number of investigations | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Kwun M Fong, Principal Investigator — UQTRC at TPCH; Steven Lam, Principal Investigator — British Columbia Cancer Agency
Locations (6):
- Australia (5):
  - St Vincent's Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- BC Cancer Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonney A, Pascoe DM, McCusker MW, Steinfort D, Marshall H, McWilliams A, Brims FJ, Stone E, Fogarty P, Silver JD, Milner B, Silverstone E, Hsu E, Nguyen D, Rofe C, White C, Hu X, Mayo J, Myers R, Fong KM, Manser R, Lam S. Incidental findings during lung low-dose computed tomography cancer screening in Australia and Canada, 2016-21: a prospective observational study. Med J Aust. 2025 May 5;222(8):403-411. doi: 10.5694/mja2.52649. PMID 40320382
- [Derived] Bonney A, Brodersen J, Siersma V, See K, Marshall HM, Steinfort D, Irving L, Lin L, Li J, Pang S, Fogarty P, Brims F, McWilliams A, Stone E, Lam S, Fong KM, Manser R. Validation of the psychosocial consequences of screening in lung cancer questionnaire in the international lung screen trial Australian cohort. Health Qual Life Outcomes. 2024 Jan 25;22(1):10. doi: 10.1186/s12955-023-02225-8. PMID 38273370
- [Derived] Cressman S, Weber MF, Ngo PJ, Wade S, Behar Harpaz S, Caruana M, Tremblay A, Manser R, Stone E, Atkar-Khattra S, Karikios D, Ho C, Fernandes A, Yi Weng J, McWilliams A, Myers R, Mayo J, Yee J, Yuan R, Marshall HM, Fong KM, Lam S, Canfell K, Tammemagi MC. Economic impact of using risk models for eligibility selection to the International lung screening Trial. Lung Cancer. 2023 Feb;176:38-45. doi: 10.1016/j.lungcan.2022.12.011. Epub 2022 Dec 22. PMID 36592498
- [Derived] Tammemagi MC, Ruparel M, Tremblay A, Myers R, Mayo J, Yee J, Atkar-Khattra S, Yuan R, Cressman S, English J, Bedard E, MacEachern P, Burrowes P, Quaife SL, Marshall H, Yang I, Bowman R, Passmore L, McWilliams A, Brims F, Lim KP, Mo L, Melsom S, Saffar B, Teh M, Sheehan R, Kuok Y, Manser R, Irving L, Steinfort D, McCusker M, Pascoe D, Fogarty P, Stone E, Lam DCL, Ng MY, Vardhanabhuti V, Berg CD, Hung RJ, Janes SM, Fong K, Lam S. USPSTF2013 versus PLCOm2012 lung cancer screening eligibility criteria (International Lung Screening Trial): interim analysis of a prospective cohort study. Lancet Oncol. 2022 Jan;23(1):138-148. doi: 10.1016/S1470-2045(21)00590-8. Epub 2021 Dec 11. PMID 34902336
- [Derived] Lim KP, Marshall H, Tammemagi M, Brims F, McWilliams A, Stone E, Manser R, Canfell K, Weber M, Connelly L, Bowman RV, Yang IA, Fogarty P, Mayo J, Yee J, Myers R, Atkar-Khattra S, Lam DCL, Rosell A, Berg CD, Fong KM, Lam S; ILST (International Lung Screening Trial) Investigator Consortium. Protocol and Rationale for the International Lung Screening Trial. Ann Am Thorac Soc. 2020 Apr;17(4):503-512. doi: 10.1513/AnnalsATS.201902-102OC. PMID 32011914